CLINICAL TRIAL: NCT00708149
Title: Phase IV Study of Comparison of the Efficacy for Stress Ulcer Prophylaxis Between the Patients Received Lansoprazole OD and Control Group Weaning From Mechanical Ventilator in Respiratory Care Center: a Randomized Control Trial
Brief Title: Comparison of the Efficacy for Stress Ulcer Prophylaxis Between the Patients Received Lansoprazole OD and Control Group Weaning From Mechanical Ventilator in Respiratory Care Center: a Randomized Control Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCLin
Record Dates: First submitted 2008-03-03; First posted 2008-07-02 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Respiratory Failure
Keywords: lansoprazole, weaning,stress ulcer prophylaxis
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): lansprazole 30 mg qd from NG route or orally
  Interventions: Drug: lansoprazole OD
- 2 (Placebo Comparator): control group without any PPI, H2 blockers or other medications for treating peptic ulcers.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lansoprazole OD — arm 1: lansprazole 30 mg qd from NG route or orally for 14 days
  Other Names: Takepron OD for PO QD
  Arms: 1
Drug: placebo — takepron placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether lansoprazole administered nasogastrically is effective for stress ulcer prophylaxis in respiratory intensive care unit.

DETAILED DESCRIPTION:
Although stress ulcer is a complication that can cause mortality and morbidity in critical patients, there is still lack of consensus about its prophylaxis. There is also few data available from Taiwan. H2 blockers are commonly used due to convenience. Some prefer sucralfate (a mucosal protective agent) for the sake of less associated nosocomial pneumonia. Recently, proton pump inhibitors were shown to have good prophylactic effects for stress ulcer. Lansoprazole has good acid suppression effect and the tablets are soluble for the use of tube feeding. There was no data about the prophylaxis of stress ulcer development during the program of weaning from the mechanical ventilators. Therefore, we conduct a study of the comparison of lansoprazole administered nasogastrically and control group for stress ulcer prophylaxis in respiratory intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Initial ICU admission, APACHE II score ≥25。
2. Evidence of IICP ( ICP monitor proved or brain CT proved edema)。
3. Evidence of peptic ulcer disease ( A or H) proved by PES more than 3 months ago without PPI or H2 blocker agents therapy in recent one week。
4. UGI bleeding history in ICU before transferring to RCC (proved by NG aspirate coffee ground substance or fresh blood ≥ 60 ml)。Not received PPI or H2 blocker agents in recent one week.
5. Received NSAID for more than 7 days。
6. Bleeding tendency or with major disease patients: coagulopathy, ESRD (CCR<10), hematologic malignancy, liver cirrhosis Child C。

Exclusion Criteria:

1. Age < 18 y/o, pregnancy。
2. Active UGI bleeding and under PPI or H2-blockers。
3. Family unwillings。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Overt UGI bleeding: (1)tarry stool or coffee ground substance or fresh blood from NG≥ 60ml (2)blood component transfusion for more than PRBC 2 units 3)PES or TAE or surgical intervention for hemostasis | The first 30 days after RCC admission

SECONDARY OUTCOMES:
30 days mortality rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Chu C Lin, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Cook DJ, Fuller HD, Guyatt GH, Marshall JC, Leasa D, Hall R, Winton TL, Rutledge F, Todd TJ, Roy P, et al. Risk factors for gastrointestinal bleeding in critically ill patients. Canadian Critical Care Trials Group. N Engl J Med. 1994 Feb 10;330(6):377-81. doi: 10.1056/NEJM199402103300601. PMID 8284001
- [Background] Daley RJ, Rebuck JA, Welage LS, Rogers FB. Prevention of stress ulceration: current trends in critical care. Crit Care Med. 2004 Oct;32(10):2008-13. doi: 10.1097/01.ccm.0000142398.73762.20. PMID 15483408
- [Background] Lam NP, Le PD, Crawford SY, Patel S. National survey of stress ulcer prophylaxis. Crit Care Med. 1999 Jan;27(1):98-103. doi: 10.1097/00003246-199901000-00034. PMID 9934901
- [Background] Tryba M, Cook D. Current guidelines on stress ulcer prophylaxis. Drugs. 1997 Oct;54(4):581-96. doi: 10.2165/00003495-199754040-00005. PMID 9339962
- [Background] Chun AH, Shi HH, Achari R, Dennis S, Cavanaugh JH. Lansoprazole: administration of the contents of a capsule dosage formulation through a nasogastric tube. Clin Ther. 1996 Sep-Oct;18(5):833-42. doi: 10.1016/s0149-2918(96)80043-9. PMID 8930427
- See also: Related Info — http://www.e-pharm.info/index.php?option=com_content&view=category&id=38&Itemid=103